CLINICAL TRIAL: NCT06454474
Title: Individualized Neuromodulation Intervention Techniques for the Core Clinical Features of Drug Addiction
Brief Title: Closed-loop tACS Modulation for the Core Clinical Features of Drug Addiction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MZhao-016
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2024-06

CONDITIONS: Amphetamine Use Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Closed-loop tACS stimulation based on addiction-induced states (Experimental): In the initial phase of this study, participants will be subjected to individual closed-loop tACS interventions for ten-days intervals. Concurrently, they will be exposed to MA-related cue paradigms to induce brain addiction states, while scalp EEG signals are collected. Stimulation will be initiated only upon identifying specific neural signals associated with MA cues.
  Interventions: Device: Closed-loop tACS stimulation based on addiction-induced states

INTERVENTIONS:
Device: Closed-loop tACS stimulation based on addiction-induced states — We conducted a longitudinal controlled study of closed-loop tACS interventions among MA dependents.This involved implementing interventions based on addiction-induced states.

SUMMARY:
Using specific EEG biomarkers in methamphetamine-dependent individuals, this study systematically probes the effect of closed-loop tACS based on brain states

DETAILED DESCRIPTION:
Methamphetamine use disorder (MUD) addiction represents a severe public health concern. Individuals addicted to methamphetamine exhibit intense cravings and physiological reactions when exposed to addiction-related cues, a phenomenon termed "cue reactivity." Cue reactivity is a critical factor in the development and persistence of addiction. Impairments in inhibitory control are considered a significant factor contributing to the emergence of cue reactivity. Conventional pharmacological and physical interventions suffer from low efficiency and high effect variance. Closed-loop physical interventions, which adjust stimulation parameters in real-time based on brain state, are an innovative approach with the potential to enhance the precision and efficiency of treatments. Closed-loop interventions based on transcranial alternating current stimulation (tACS) hold promise as a novel therapeutic method for treating methamphetamine addiction. This study aims to develop and evaluate the effect of closed-loop tACS on cue reactivity and inhibition control function in MUD. Therefore, the investigators intend to employ the non-invasive tACS technique, predicated upon biomarkers of addiction states, to administer specific frequency stimulations to targeted brain regions, aiming to achieve therapeutic objectives in addiction treatment.

ELIGIBILITY:
Inclusion Criteria:

Individuals aged between 18 and 45 years, irrespective of gender, having completed a minimum of 9 years of education and capable of effectively cooperating in questionnaire evaluations.

Meet the diagnostic criteria set forth by the DSM-V concerning the severity of amphetamine-type substance addiction.

A history of utilizing amphetamine-type substances for a duration not less than one year, with a frequency of use being at least once per week.

Consent to actively cooperate in the completion of subsequent follow-up assessments.

Exclusion Criteria:

Severe cognitive functional impairments manifested through a history of head trauma, cerebrovascular diseases, epilepsy, etc., or usage of cognitive enhancement drugs in the past 6 months; an intellectual disability with an IQ score less than 70.

A diagnosis of schizophrenia or other severe mental illnesses as per the DSM-5 criteria.

Abuse or dependence on other psychoactive substances (excluding nicotine) within the past 5 years.

Severe organic diseases that might compromise study participation. Contraindications to tACS, such as a history of epileptic seizures or the presence of metallic implants in proximity to the head.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2024-06-30 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Change of Craving assessed by Visual Analog Scale (VAS) | through study completion, an average of 1 month
  The intensity of psychological craving in MA dependents was assessed using the Visual Analogue Scale (VAS), where individuals rated their cravings on a scale from 0 to 10, with higher scores indicating greater levels of craving. The VAS scores were utilized based on two conditions: during a resting state and when subjected to cue induction involving images associated with methamphetamine, serving as the criteria for evaluation.

SECONDARY OUTCOMES:
Stop-signal task | through study completion, an average of 1 monoth
  The stop-signal task can indicate executive control capabilities by measuring Stop-signal reaction time, Stop-signal delays, Go-task reaction time, and Success and failure inhibition rates.
Drug Use | through study completion, an average of 1 month
  OCDUSE scale

CONTACTS AND LOCATIONS:
Overall Officials: MIn Zhao, Study Chair — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai, Shanghai, China, 200000, China

IPD SHARING:
Plan to Share IPD: No